CLINICAL TRIAL: NCT01441674
Title: The Effectiveness of Animal Assisted Therapy for Children Hospitalized in a Pediatric Setting
Brief Title: Animal Assisted Therapy in a Pediatric Setting
Acronym: AAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AAT-IRB#1011-089
Record Dates: First submitted 2011-01-28; First posted 2011-09-28 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Developmental Delays; Global Developmental Delay; Stroke; Cancers; Seizures Disorders; Behavior Problems; Feeding Disorder; Developmental Delay in Feeding
Keywords: Occupational Therapy
MeSH Terms: conditions — Learning Disabilities; Stroke; Neoplasms; Mental Disorders; Feeding and Eating Disorders | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Animal Assisted Therapy Visit 1 (Experimental): Standard OT Therapy with Animal Assisted Therapy at Visit 1 and Not at Visit 2
  Interventions: Behavioral: Animal Assisted Therapy
- Animal Assisted Therapy at Visit 2 (Experimental): Standard OT Therapy with Animal Assisted Therapy at Visit 2 and not Visit 1
  Interventions: Behavioral: Animal Assisted Therapy

INTERVENTIONS:
Behavioral: Animal Assisted Therapy — There will be a therapy dog and dog trainer present working with the patient for the AAT arm.
  Other Names: Group 1 and Group 2

SUMMARY:
The primary purpose for this study is to determine if children who receive Occupational Therapy while they are an inpatient in the hospital will be more motivated to participate in therapy as well as increase the amount of time they will work during that particular session when a therapy dog is present during their sessions. The investigators will also be collecting data regarding a child's heart rate and blood pressure prior to the session starting and ending to determine if having a therapy dog present also helps relax a child.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate if a patient in the pediatric acute care setting receiving Occupational Therapy (OT) services in adjunct with animal assisted therapy (AAT) are more motivated to actively participate in the therapy session for a longer period of time.

Methods:

Thirty inpatients will be recruited to participate in this study. This study will utilize a randomized crossover study design where the patients act as their own control. The treatment period for hospitalized patients will include an on off pattern of incorporating AAT into their OT session. Patients' participation of therapy will be assessed with a participation scale (see Figure 2) and the OT session time. Patients will be evaluated for OT and the therapist will determine goals based on functional status and needs of the particular patient. Goals will be determined by providing a functional evaluation based upon Occupational Therapists clinical observation, developmental standards and current functional level of the patient.

Patients who are potential candidates for this study will be hospitalized at Children's Hospitals and Clinics of Minnesota on the St. Paul campus. All inpatients stated to have decreased functional skills that have been referred by a physician to OT will be invited to participate this study.

Patients have a difficult time participating in various therapies due to emotional stress, anxiety, and feeling uncomfortable with the hospital environment. Limited studies have demonstrated the value of AAT used in conjunction with OT for children, regardless of diagnosis within the hospital setting. Results of this study can justify the use of this valuable therapy not only for the selected population, but also for other disciplines such as physical and speech therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient Occupational Therapy Referrals
* Ages 0-21 years

Exclusion Criteria:

* Patients who are uncomfortable with dogs
* Patients who exhibits violent behavior
* Animal Allergies
* Patients are unable to work with a dog
* Patients who exhibit severe cognitive delays

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
OT Participation scale | 4 days
  The patients response to therapy can be measures using the following behavior domains (cognition, fine motor, activities and daily living, feeding skills, active range of motion/activities, and functional Transfers).

SECONDARY OUTCOMES:
Vital Signs (Blood Pressure and heart rate) | 4 days
  Heart rate and blood pressure will be measured to assess if AAT minimizes stress and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Iammatteo, OT, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hopsitals and Clinics of Minnesota, Saint Paul, Minnesota, United States